CLINICAL TRIAL: NCT00621686
Title: Phase II Trial of Bevacizumab in Combination With Sorafenib in Recurrent Glioblastoma Multiforme
Brief Title: Bevacizumab and Sorafenib in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0776; NCI-2009-00832 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000587614 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-02-21; First posted 2008-02-22 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Bevacizumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib + Bevacizumab/Group A (Experimental): Patients receive oral sorafenib 400 mg (200 mg twice daily) days 1-5 and 8-12 and 5 mg/kg bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 14 days.
  Patients undergo blood and plasma sample collection at baseline and then periodically during study treatment for translational research studies. Translational research studies include analysis of circulating endothelial cells and circulating endothelial progenitor cells by flow cytometry and measurement of angiogenic proteins in plasma by ELISA. DNA and buffy coat are extracted and collected from the blood samples for pharmacogenetic studies.
  Quality of life is assessed at baseline, prior to every other treatment course, and at the end of treatment.
  After completion of study treatment, patients are followed at 28-42 days, every 3 months for 5 years, and then annually for 10 years.
  Interventions: Biological: bevacizumab; Drug: sorafenib tosylate
- Sorafenib + Bevacizumab /Group B (Experimental): Patients receive oral sorafenib 200 mg once daily on days 1-14 and 5 mg/kg bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 14 days.
  Patients undergo blood and plasma sample collection at baseline and then periodically during study treatment for translational research studies. Translational research studies include analysis of circulating endothelial cells and circulating endothelial progenitor cells by flow cytometry and measurement of angiogenic proteins in plasma by ELISA. DNA and buffy coat are extracted and collected from the blood samples for pharmacogenetic studies.
  Quality of life is assessed at baseline, prior to every other treatment course, and at the end of treatment.
  After completion of study treatment, patients are followed at 28-42 days, every 3 months for 5 years, and then annually for 10 years.
  Interventions: Biological: bevacizumab; Drug: sorafenib tosylate

INTERVENTIONS:
Biological: bevacizumab
Drug: sorafenib tosylate

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab and sorafenib may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving bevacizumab together with sorafenib may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving bevacizumab together with sorafenib works in treating patients with recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify the clinical efficacy of bevacizumab and sorafenib, as measured by 6-month progression-free survival, in patients with recurrent glioblastoma multiforme.

Secondary

* Assess time to progression of this patient population.
* Assess overall survival of this patient population.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib once daily on days 1-14 and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood and plasma sample collection at baseline and then periodically during study treatment for translational research studies. Translational research studies include analysis of circulating endothelial cells and circulating endothelial progenitor cells by flow cytometry and measurement of angiogenic proteins in plasma by ELISA. DNA and buffy coat are extracted and collected from the blood samples for pharmacogenetic studies.

Quality of life is assessed at baseline, prior to every other treatment course, and at the end of treatment.

After completion of study treatment, patients are followed at 28-42 days, every 3 months for 5 years, and then annually for 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme as determined by pre-registration central pathology review

  * Gliosarcoma allowed
* Must have evidence of tumor progression by MRI or CT scan following radiotherapy or the most recent anti-tumor therapy
* No more than 1 chemotherapy regimen for progressive or recurrent disease
* Bidimensionally measurable or evaluable disease by MRI or CT scan
* No evidence of CNS hemorrhage on baseline CT or MRI

  * Patients with T1 hyperintensity confined to the surgical cavity which is felt likely due to post surgical blood contaminating the intracavity cerebrospinal fluid or irrigation that have not yet absorbed and which is not felt to clinically or radiographically represent new spontaneous hemorrhage are eligible
  * Patients with old blood products or hemosiderin without a history of spontaneous bleeding are eligible

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin > 9.0 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal
* AST ≤ 3 times upper limit of normal
* Creatinine ≤ upper limit of normal
* Urine protein:creatinine ratio < 1 OR urine protein < 1,000 mg by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for six months after completion of study treatment
* Able to complete questionnaire(s) alone or with assistance
* Willing to return to NCCTG enrolling institution for follow-up
* Willing to provide mandatory blood samples for research purposes
* Not immunocompromised (other than that related to the use of corticosteroids)
* No known HIV positivity
* No concurrent uncontrolled illness including, but not limited to, the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* No inadequately controlled hypertension (i.e., systolic blood pressure [BP] > 150 mm Hg or diastolic BP > 100 mm Hg while on antihypertensive medications)

  * Patients with well-controlled hypertension are eligible
* No myocardial infarction or unstable angina within the past 6 months
* No congestive heart failure requiring the use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* No New York Heart Association class II-IV congestive heart failure
* No significant vascular disease (e.g., aortic aneurysm or aortic dissection)
* No peripheral arterial thrombosis within the past 6 months
* No stroke or transient ischemic attack within the past 6 months
* No history of hypertensive crisis or hypertensive encephalopathy
* No evidence of bleeding diathesis (greater than normal risk of bleeding) or coagulopathy (in the absence of therapeutic anticoagulation)
* No active or recent history of hemoptysis (i.e., ≥ ½ teaspoon of bright red blood per episode) within the past 30 days
* No serious, nonhealing wounds, ulcers, or bone fractures
* No condition that impairs the ability to swallow pills (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation)
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No significant traumatic injury within the past 28 days
* No known hypersensitivity to any of the components of sorafenib or bevacizumab
* No other active malignancy within the past 3 years, except nonmelanoma skin cancer or carcinoma in situ of the cervix

  * Patients with a history of prior malignancy must not be receiving specific treatment (other than hormonal therapy) for that malignancy
* No co-morbid systemic illness or other concurrent severe disease that, in the judgment of the investigator, would make the patient inappropriate for entry into this study or significantly interfere with the proper assessment of safety and toxicity of the prescribed study regimen

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 12 weeks since prior radiotherapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* More than 2 weeks since prior small molecule cell cycle inhibitors
* At least 1 week since prior fixed-dose corticosteroids (or no corticosteroids)
* No prior intratumoral chemotherapy, stereotactic radiosurgery or interstitial brachytherapy unless there is a separate lesion on MRI that is not part of the prior treatment field OR there is proof of recurrent disease based on biopsy, MRI spectroscopy, or PET scan
* No prior antiangiogenic therapy
* No prior surgical procedures affecting absorption
* More than 7 days since prior core biopsy or other minor surgical procedures

  * Placement of a vascular access device is allowed
* More than 28 days since prior major surgical procedure or open biopsy
* No concurrent major surgical procedure
* No other concurrent investigational agents
* No concurrent enzyme-inducing antiepileptic drugs (e.g., phenytoin, fosphenytoin, carbamazepine, phenobarbital, or primidone)
* No other concurrent potent CYP3A4 inducers (e.g., rifampin or St. John's wort)
* No concurrent therapeutic anticoagulation with warfarin

  * Prophylactic anticoagulation (i.e., low-dose warfarin) for venous or arterial access devices allowed provided the INR < 1.5
  * Therapeutic anticoagulation with low molecular weight heparin allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2014-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, MD, Study Chair — Mayo Clinic
Locations (204):
- United States (204):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Cancer Care Associates, Fresno, California
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Drs. Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Northwest Cancer Specialists at Rose Quarter Cancer Center, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Luther Midlelfort Hospital, Eau Claire, Wisconsin
  - Midelfort Clinic - Luther, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Galanis E, Jaeckle KA, Anderson S, et al.: NCCTG phase II trial of bevacizumab in combination with sorafenib in recurrent GBM. [Abstract] J Clin Oncol 28 (Suppl 15): A-2018, 2010.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib + Bevacizumab/Group A: Patients receive oral sorafenib 400 mg (200 mg twice daily) days 1-5 and 8-12 and 5 mg/kg bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 14 days.
- Sorafenib + Bevacizumab /Group B: Patients receive oral sorafenib 200 mg once daily on days 1-14 and 5 mg/kg bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 14 days.
Period: Overall Study
Arm/Group | Sorafenib + Bevacizumab/Group A | Sorafenib + Bevacizumab /Group B
Started | 19 | 35
Completed | 19 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib + Bevacizumab/Group A | Sorafenib + Bevacizumab /Group B | Total
Number analyzed (Participants) | 19 | 35 | 54
Age, Continuous [Median (Full Range); unit: years] | 54 [25 to 68] | 55 [28 to 76] | 55 [25 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 12 | 23 | 35
Region of Enrollment [Number; unit: participants]
  United States | 19 | 35 | 54

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival
Description: Primary Endpoint: 6-month progression free survival (PFS6): The proportion of successes will be estimated using the binomial point estimator (number of successes divided by the total number of evaluable patients) and the binomial 95% confidence interval estimated. To be classified as a success, an evaluable patient must be alive and progression-free 6 months after registration to the study. Patients who die prior to 6 months after study registration will be considered to have failed. Progression is defined as a >25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions or unequivocal increase in size of contrast enhancement or increase in mass effect as agreed upon independently by primary physician and quality control physicians: appearance of new lesions compared to pretreatment MRI and/or CT scan.
Time Frame: at 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Sorafenib + Bevacizumab /Group B: Patients receive oral sorafenib 200 mg once daily on days 1-14 and 5mg/kg bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 14 days.
Arm/Group | Sorafenib + Bevacizumab/Group A | Sorafenib + Bevacizumab /Group B
Number analyzed (Participants) | 19 | 35
proportion of participants | 0.263 [0.101 to 0.514] | 0.171 [0.072 to 0.343]

2. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) is defined to be the length of time from study registration to a) date of disease progression as defined by section 11.0 of the protocol, or b) last follow-up. If a patient dies without documentation of disease progression, the patient will be considered to have had a tumor progression at the time of death unless there is sufficient documented evidence to conclude no progression occurred prior to death. Time to progression curves were compared via the log-rank test. Progression is defined as a >25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions or unequivocal increase in size of contrast enhancement or increase in mass effect as agreed upon independently by primary physician and quality control physicians: appearance of new lesions compared to pretreatment MRI and/or CT scan.
Time Frame: Time from study registration to a) date of disease progression, or b) last follow-up; Up to 15 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib + Bevacizumab/Group A | Sorafenib + Bevacizumab /Group B
Number analyzed (Participants) | 19 | 35
months | 3.61 [1.84 to 5.95] | 2.66 [2.07 to 3.25]
Statistical Analysis 1: Comparison: Sorafenib + Bevacizumab/Group A vs Sorafenib + Bevacizumab /Group B; Test type: Superiority or Other; p = 0.069, Log Rank

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the length of time from date of registration to a) date of death due to any cause or b) last follow-up.
Time Frame: Time from date of registration to a) date of death due to any cause or b) last follow-up; Up to 15 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib + Bevacizumab/Group A | Sorafenib + Bevacizumab /Group B
Number analyzed (Participants) | 19 | 35
months | 5.58 [4.11 to 8.48] | 5.62 [3.22 to 8.67]

ADVERSE EVENTS:
Time Frame: Adverse event assessments were collected ≤21 days prior to registration, prior to each new treatment cycle, at PD, withdrawal, or removal, and 28-42 days after treatment discontinuation; for up to 2 years.
Description: This study will utilize the Common Terminology Criteria for Adverse Events (CTCAE) v3.0 for adverse event monitoring and reporting. The CTCAE v3.0 can be accessed from the CTEP home page http://ctep.cancer.gov.
Arm/Group | Sorafenib + Bevacizumab/Group A | Sorafenib + Bevacizumab /Group B
Serious Adverse Events (participants affected / at risk) | 9/19 | 9/35
Other Adverse Events (participants affected / at risk) | 19/19 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib + Bevacizumab/Group A (N=19) | Sorafenib + Bevacizumab /Group B (N=35)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (3) | 3 (4)
Fever (General disorders) | 0 (0) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 3 (4) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib + Bevacizumab/Group A (N=19) | Sorafenib + Bevacizumab /Group B (N=35)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (25) | 16 (26)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 9 (22) | 11 (24)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 7 (11) | 8 (20)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 5 (6) | 8 (18)
Nausea (Gastrointestinal disorders) | 7 (15) | 13 (22)
Oral pain (Gastrointestinal disorders) | 1 (3) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5) | 5 (6)
Disease progression (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (3) | 1 (2)
Fatigue (General disorders) | 18 (118) | 34 (220)
Fever (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 3 (6)
Alanine aminotransferase increased (Investigations) | 2 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Bilirubin increased (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 4 (10) | 9 (14)
Lipase increased (Investigations) | 3 (3) | 3 (5)
Lymphocyte count decreased (Investigations) | 3 (6) | 13 (29)
Neutrophil count decreased (Investigations) | 2 (3) | 1 (3)
Platelet count decreased (Investigations) | 10 (52) | 17 (31)
Weight loss (Investigations) | 5 (39) | 10 (30)
Anorexia (Metabolism and nutrition disorders) | 8 (22) | 10 (26)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 6 (10) | 7 (13)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Abducens nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 2 (3) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (11) | 3 (5)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 4 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (5)
Seizure (Nervous system disorders) | 0 (0) | 5 (5)
Speech disorder (Nervous system disorders) | 1 (4) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 2 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (5)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (9)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (11)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 7 (40) | 12 (30)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 7 (14) | 12 (29)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 9 (22) | 25 (84)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes